CLINICAL TRIAL: NCT02188771
Title: A Phase I, Prospective, Randomized, Open-label, Active-Controlled Clinical Trial for Safety Evaluation of Intra-articular Injection of RegenoGel-SP for the Treatment of Moderate to Severe Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ProCore Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROC- 1
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2014-07

CONDITIONS: Osteoarthritis
Keywords: Moderate to Severe OA; VAS score of ≥ 5; grade III-IV Kellgren Lawrence of OA; subjects who failed conservative treatment; subjects who candidates for total knee replacement (TKR); subject 45 and 75 years old; subject is experiencing pain in the intended study knee with a VAS score of ≥ 5; subject has a Body Mass Index (BMI) between 18.5 and 35
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RegenoGel SP 2ml (Experimental): RegenoGel-SP is a new viscosupplement intended for the intra-articular treatment of OA.
  Following signing the Informed Consent form (Visit 1), subjects who conform to the inclusion criteria will be evaluated for vital signs, blood hematology, chemistry, INR, aPTT and ECG, and will be subjected to a 30-40ml blood withdrawal that will be used for the production of autologous RegenoGel-SP. Subjects randomized to receive RegenoGel-SP will receive a single, intra-articular injection (Visit 2).
  Interventions: Device: intra-articular administration of RegenoGel-SP or hyaluronic acid (HA)

INTERVENTIONS:
Device: intra-articular administration of RegenoGel-SP or hyaluronic acid (HA) — Intra-articular Injection: single injection of RegenoGel SP or 3 injections of HA

SUMMARY:
This is a Phase I, prospective, active-controlled, randomized, open-label, clinical trial designed to assess the safety and tolerability of single intra-articular injection of RegenoGel-SP for the treatment of OA.

RegenoGel-SP is composed of fibrinogen in plasma linked to a high molecular weight HA. The viscoelastic properties resulting from the combination of these two natural macromolecules is further enhanced by joint surface associated factors to generate a viscoelastic gel with superior stability and mechanical integrity.

DETAILED DESCRIPTION:
Eighteen subjects will be randomized and sequentially assigned to RegenoGel-SP or to hyaluronic acid (HA) treatments on a 2:1 basis, respectively. Treatment groups will be assigned as per a randomization list that will be prepared prior to the start of the study. Randomization will be done at Enrollment (Visit 2). Neither surgeon nor subject will be blinded to treatment. Subjects will be monitored for 6 months following treatment. Following signing the Informed Consent form (Visit 1), subjects who conform to the inclusion criteria will answer questionnaires for grading of their symptoms, pain level and overall functional performance. Subjects will be evaluated for vital signs, blood hematology, chemistry, INR, aPTT and ECG, and will be subjected to a 30-40ml blood withdrawal that will be used for the production of autologous RegenoGel-SP. Subjects randomized to receive RegenoGel-SP will receive a single, intra-articular injection (Visit 2), while subjects randomized to receive HA treatment (Euflexxa®) will be injected with 3 intra-articular weekly injections of (Visits 2-4). Subjects treated with RegenoGel-SP will attend visits 3 and 4 but will not receive treatment. All subjects will return for Observation visits after 6 weeks, 3 months and 6 months following treatment (Visits 5-7). During treatment and observation visits, subjects will be monitored for safety parameters (local and systemic AEs, blood work analysis ) and response to treatment using the above questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated the informed consent form
* Subject is experiencing pain in the intended study knee with a VAS score of ≥ 5
* Subject with degenerative changes in the intended study knee that can be categorized as grade III-IV Kellgren Lawrence based upon standing posterior-anterior and lateral radiographs of the knee and is a candidate for TKR
* Subject has a Body Mass Index (BMI) between 18.5 and 35
* Subject has failed conservative treatments to the intended study knee, including such measures as weight reduction, physical therapy, hydrotherapy, analgesics, non-steroidal anti-inflammatory drugs (NSAIDs) and/or intra-articular injections

Exclusion Criteria:

* Subjects with history of significant knee trauma to the intended study knee or with previous arthroscopic surgery of the intended study knee within the last 3 months preceding screening
* Subject had any intra-articular injections to the intended study knee within 6 months prior to Screening
* Subject is unable to stop chronic administration of pain medications (including paracetamol), from the day before each study visit through completion of the study visit.
* Subject has a history of Psoriatic Arthritis, Rheumatoid Arthritis,or any other inflammatory condition associated with arthritis
* Subject has a superficial wound in the area of the intended study knee
* Subject has known sensitivity to any of the treatment components, egg, rubber or latex
* Subject has a history of anaphylactic shock or other severe systemic response or other adverse event to human blood products
* Subject has a clinically significant abnormal finding (e.g., laboratory result or ECG) on screening
* Subject has clinically significant abnormal INR or aPTT coagulation result.
* Subject has a hemoglobin concentration below 10.5
* Subject is positive for Human Immunodeficiency Virus / Aquired Immunodeficiency Syndrome (HIV/AIDS), Hepatitis B or C viral infections, or acute or chronic liver disease
* Subject has ever had cellulitis of the lower extremities, a superficial or deep vein thrombosis, or a family history of a clotting disorders
* Subject has had cancer in the past 5 years or surgery involving the chest, abdomen, pelvis, or lower extremities in the past year
* Subject receives any investigational device or product within 30 days of Visit l
* Subject has any recent (acute) or chronic medical, psychiatric, or social problem that might: 1) interfere with the Subject's performance or completion of the trial; 2) obfuscate the Subject's study data; or 3) render the Subject unable to understand the nature, scope, and possible consequences of the study
* Subject is receiving an oral or injected anticoagulant
* Subject ever abused drugs or alcohol (self-reported)
* Subject received a blood transfusion within 6 months prior to Visit 1.
* Subject donated blood or blood products within 3 months prior to Visit 1.
* Subject has any elective surgery of any kind to the lower extremities or elective surgery requiring general anesthesia scheduled during the course of the trial

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Clinical safety and tolerability | 6 month following RegenoGel injection
  Incidence, relatedness, and severity of treatment-emergent SAEs, UAEs, AEs in the 2 treatment arms.
  Supportive safety measures:
  * Local safety outcomes (presence of erythema, edema, swelling, effusion, pain, sensitivity in the treated knee)
  * Global clinical assessment
  * Pain assessment
  * Percentage of subjects who discontinued the study due to AEs
  * Laboratory tests (haematology, blood chemistry, INR, aPTT), ECG and vital signs

SECONDARY OUTCOMES:
Efficacy assessment | 6 month following RegenoGel injection
  * Change in pain in the affected knee joint in response to treatments using the Visual Analog Score (VAS).
  * Change in the subject´s activity in response to treatments based on the WOMAC evaluation form.
  * Change in quality of life at baseline in response to treatments using the SF-36v2 health survey.
  * Change in joint space width using standard X-ray in response to treatments

CONTACTS AND LOCATIONS:
Overall Officials: Gabrilet Agar, Dr, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Zrifin, Israel